CLINICAL TRIAL: NCT00120705
Title: A Randomized, Open-Label, Pilot Study to Evaluate Every Three Week Maintenance Dosing of Darbepoetin Alfa Therapy in Anemic Subjects With Non-Myeloid Malignancies Receiving Chemotherapy
Brief Title: Treatment for Anemic Subjects With Non-Myeloid Malignancies Receiving Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20020167
Record Dates: First submitted 2005-06-30; First posted 2005-07-19 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Neoplasms; Anemia
Keywords: anemia; darbepoetin alfa; Amgen; Non-myeloid Malignancies
MeSH Terms: conditions — Neoplasms; Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa

SUMMARY:
The purpose of this study is to assess the ability of darbepoetin alfa to maintain hemoglobin concentrations greater than or equal to 10 g/dL when administered every 3 weeks (Q3W).

ELIGIBILITY:
Inclusion Criteria: - Subjects with non-myeloid malignancies - Anemia (screening hemoglobin concentration greater than or equal to 10.5 g/dL but less than or equal to 12.0 g/dL) related to cancer and chemotherapy - At least 8 additional weeks of cyclic chemotherapy planned regardless of schedule - Karnofsky Performance Status of greater than or equal to 50% - Serum creatinine concentration less than or equal to 2.0 mg/dL Exclusion Criteria: - Iron deficiency - Red blood cell (RBC) transfusion within 4 weeks of screening - Unstable cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204
Dates: Start 2002-11; Study Completion 2003-09

PRIMARY OUTCOMES:
To assess the ability of darbepoetin alfa to maintain hemoglobin concentrations greater than or equal to 10 g/dL when administered every 3 weeks (Q3W)

SECONDARY OUTCOMES:
Assess safety profile of subjects treated with darbepoetin alfa

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Charu V, Saidman B, Ben-Jacob A, Justice GR, Maniam AS, Tomita D, Rossi G, Rearden T, Glaspy J. A randomized, open-label, multicenter trial of immediate versus delayed intervention with darbepoetin alfa for chemotherapy-induced anemia. Oncologist. 2007 Oct;12(10):1253-63. doi: 10.1634/theoncologist.12-10-1253. PMID 17962619
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com